CLINICAL TRIAL: NCT01036022
Title: A Double-Blind, Double-Dummy, Placebo- and Active-Controlled Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Anti-Inflammatory Effects of GSK1399686 in Patients With Mild to Moderately Active Ulcerative Colitis
Brief Title: Effect of GSK1399686 in Patients With Mild to Moderately Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 111407
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Colitis, Ulcerative
Keywords: mesalazine; ulcerative colitis; pharmacokinetics/dynamics; GSK1399686
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 2 (Experimental): ASACOL 800mg t.i.d.
  Interventions: Drug: GSK1399686
- Group 1 (Experimental): GSK1399686 at 3-4 dose levels
  Interventions: Drug: GSK1399686
- Group 3 (Experimental): Placebo
  Interventions: Drug: GSK1399686

INTERVENTIONS:
Drug: GSK1399686 — Each dose level of GSK1399686 will be subsequently tested in a cohort of approximately 20 patients, who will be randomized in a 3:1:1 ratio to receive GSK1399686 (once daily over 4 weeks, followed by 2 weeks dosing with placebo), placebo, or ASACOL (t.i.d. for 6 weeks), respectively.

SUMMARY:
This study is the first-time-in-patient trial of GSK1399686, a novel locally-acting anti-inflammatory compound, aimed at obtaining initial information on the tolerability, safety, pharmacokinetics (including concentrations in colon mucosa) and anti-inflammatory activity of GSK1399686 upon oral dosing in patients with active ulcerative colitis.

The study is designed as a randomized, double-blind, double-dummy, placebo-controlled, sequential dose escalating trial, with an active control (ASACOL) group as internal control. Up to three cohorts (Cohorts 1-3), each consisting of approximately 20 patients with mild-moderately active ulcerative colitis not limited to the rectum, will be included, one for each dose level of GSK1399686 to be tested. Within a cohort, patients will be randomized in a 3:1:1 ratio to receive GSK1399686 (once daily over 4 weeks, followed by 2 weeks dosing with placebo), placebo, or ASACOL (t.i.d. for 6 weeks), respectively.

An interim analysis of fecal markers and disease activity data will be performed by the end of Cohort 3. Based upon results, the study may be stopped or continued by recruiting either Cohort 4 (if data on an additional dose level would be warranted to establish or clarify a dose-response relationship) or, in the case of a robust efficacy signal at any dose level previously studied, Cohort 5 (to expand the sample size for given dose level in order to evaluate the efficacy of GSK1399686). The number of patients and randomization allocation ratio may be altered in Cohort 5 and it may not include an active control arm. If Cohort 4 is initiated upon interim analysis, then a second interim analysis may be performed at the end of Cohort 4, to assess whether progression into Cohort 5 (as defined above) would be justifiable.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of non-childbearing potential between 18 and 65 years of age inclusive.
2. Presence of mild-to-moderately active ulcerative colitis spread beyond the rectum as evidenced by clinical signs and endoscopy.
3. UCDAI score 4-10 (inclusive) with rectal bleeding score ≥ 1, endoscopy score ≥ 1 and Physician's rating of disease activity < 3.
4. Body weight > or = to 50 kg and BMI within the range 18.5-29.9 kg/m2 (inclusive).
5. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

1. History of sensitivity to any component of study medications, history of hypersensitivity to ACTH, or a history of drug or other allergy that, in the opinion of the Investigator, contraindicates patient's participation in the study.
2. History of renal sensitivity to 5-ASA or presence of nephritis, nephropathia or renal function impairment.
3. Presence or a history of asthma or presence or history of other serious allergic disorder.
4. Presence or history of chronic liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
5. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
6. Presence of significant hematologic disorder, or significant bleeding or immune system disorder.
7. QTcB or QTcF >450 msec; or QTc >480 msec in patients with Bundle Branch Block, based on an average QTc value of triplicate ECGs, if the first ECG showed an abnormal value.
8. Presence of a significant cardiac, pulmonary, metabolic or infectious disease or mental disorder that, in the opinion of the Investigator, represents an unacceptable safety risk for participation in this trial.
9. History of malignant neoplastic disease within the past 5 years other than localized basal cell skin cancer, squamous cell skin cancer or cancer in situ that has been resected.
10. History of regular alcohol consumption within 6 months of the study or presence of recreational drug abuse or dependence.
11. Presence of infectious colitis as evidenced by stool culture positive for enteric pathogens or positive Clostridium difficile cytotoxin assay.
12. Suspicion of Crohn's disease, indeterminate colitis, microscopic colitis, ischaemic colitis or radiation-induced colitis, based on medical history, endoscopy and/or histological findings.
13. Bowel surgery within last 12 months.
14. Treatment with oral aminosalicylates at dose ≥ 2.4 g/day and/or with topical aminosalicylates at any dose within 2 weeks prior to Day 1 visit.
15. Treatment with systemic or topical corticosteroids within 4 weeks prior to Day 1 visit.
16. Treatment with TNF-α inhibitors or other biologics within 2 months prior to Day 1 visit.
17. Treatment with immunosuppressants (azathioprine or 6-mercaptopurine), if initiated within 3 months prior to Day 1 visit, or if changed in terms of drug or dose within 3 months prior to Day 1 visit.
18. Regular use of probiotic or prebiotic preparations, if initiated within 4 weeks prior to Day 1 visit.
19. Regular daily use of non-steroidal anti-inflammatory drugs (NSAIDs), except low dose aspirin (325 mg/day) for cardioprotection, within 7 days prior to Day 1 visit.
20. Treatment with medications known to be strong inducers of CYP3A4/5 (e.g. carbamezipine, phenobarbital, phenytoin, rifabutin, rifampin, troglitazone) or regular use of St. John's Wort within 14 days prior to Day 1 visit.
21. Treatment with medications known to be strong inhibitors of CYP3A4/5 (e.g. ketoconazole, itraconazole, fluconazole, mibefradil, clarithromycin, erythromycin, diltiazem, verapamil), or regular use of grapefruit juice within 7 days prior to Day 1 visit.
22. Treatment with medications known to be sensitive CYP3A4 substrates with a narrow therapeutic index (e.g. alfentanil, astemizole, cisapride, cyclosporine, diergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, tacrolimus, terfenadine) within 7 days prior to Day 1 visit.
23. Participation in a clinical trial and treatment with an investigational product within the following time period prior to the Day 1 visit: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
24. Prior enrolment in the present trial.

    For Canadian sites only:
25. Patients with existing gastric or duodenal ulcers.
26. Patients with urinary tract obstruction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-09-15 (Actual); Primary Completion 2013-01-10 (Actual); Study Completion 2013-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- Belgium (3):
  - GSK Investigational Site, Bonheiden
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
- Canada (5):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Vaughan, Ontario
  - GSK Investigational Site, Québec, Quebec
- Germany (9):
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Norway (3):
  - GSK Investigational Site, Lørenskog
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Tønsberg
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 111407 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111407 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111407 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111407 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111407 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111407 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111407 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 21 centres in Europe and 5 centres in Canada from 15 September 2009 to 29 July 2012.
Pre-assignment Details: A total of 78 participants with mild-moderately active ulcerative colitis not limited to the rectum were randomized in the study to receive oral dose of 4 dose levels (10 milligram [mg], 30 mg, 100 mg and 300 mg) of GSK1399686, asacol or placebo.
Groups:
- Placebo: Participants were administered oral dose of matching placebo to GSK1399686 (10 mg, 30 mg, 100 mg, 300 mg) once daily taken as 1 capsule in the morning immediately before or within 1 hour after a meal, and matching placebo to asacol taken as 1 or 2 capsules three times a day (TID) as directed by the investigator for Week 1 to Week 6. Topical 5-aminosalicylic acid (5-ASA) preparation was used as a rescue therapy.
- GSK1399686 10 mg: Participants were administered oral dose of GSK1399686 10 mg capsule once daily in the morning taken immediately before or within 1 hour after a meal for Week 1 to Week 4. Blinding was maintained by administration of matching placebo to asacol taken as 1 or 2 capsules as directed by the investigator TID for Week 1 to Week 6 and matching placebo to GSK1399686 10 mg once daily taken as 1capsule immediately before or within 1 hour after a meal in the morning for Week 5 to Week 6. Topical 5-ASA preparation was used as a rescue therapy.
- GSK1399686 30 mg: Participants were administered oral dose of GSK1399686 30 mg capsule once daily in the morning taken immediately before or within 1 hour after a meal for Week 1 to Week 4. Blinding was maintained by administration of matching placebo to asacol taken as 1 or 2 capsules as directed by the investigator TID for Week 1 to Week 6 and matching placebo to GSK1399686 30 mg once daily taken as 1capsule immediately before or within 1 hour after a meal in the morning for Week 5 to Week 6. Topical 5-ASA preparation was used as a rescue therapy.
- GSK1399686 100 mg: Participants were administered oral dose of GSK1399686 100 mg capsule once daily in the morning taken immediately before or within 1 hour after a meal for Week 1 to Week 4. Blinding was maintained by administration of matching placebo to asacol taken as 1 or 2 capsules as directed by the investigator TID for Week 1 to Week 6 and matching placebo to GSK1399686 100 mg once daily taken as 1capsule immediately before or within 1 hour after a meal in the morning for Week 5 to Week 6. Topical 5-ASA preparation was used as a rescue therapy.
- GSK1399686 300 mg: Participants were administered oral dose of GSK1399686 300 mg capsule once daily in the morning taken immediately before or within 1 hour after a meal for Week 1 to Week 4. Blinding was maintained by administration of matching placebo to asacol taken as 1 or 2 capsules as directed by the investigator TID for Week 1 to Week 6 and matching placebo to GSK1399686 300 mg once daily taken as 1capsule immediately before or within 1 hour after a meal in the morning for Week 5 to Week 6. Topical 5-ASA preparation was used as a rescue therapy.
- Asacol: Participants were administered oral dose of asacol at 400 mg or 800 mg taken as 1 or 2 capsules TID as directed by the investigator, depending on the 5-ASA dose received by the participants for Week 1 to Week 6. Blinding was maintained by administration of matching placebo to GSK1399686 (10 mg, 30 mg, 100 mg, 300 mg) once daily taken as 1capsule immediately before or within 1 hour after a meal in the morning for Week 1 to Week 6. Topical 5-ASA preparation was used as a rescue therapy.
Period: Overall Study
Arm/Group | Placebo | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg | Asacol
Started | 15 | 11 | 12 | 12 | 12 | 16
Completed | 13 | 7 | 8 | 10 | 9 | 13
Not Completed | 2 | 4 | 4 | 2 | 3 | 3
Not completed — Adverse Event | 1 | 3 | 2 | 1 | 0 | 2
Not completed — Lack of Efficacy | 1 | 1 | 1 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants were administered oral dose of matching placebo to GSK1399686 (10 mg, 30 mg, 100 mg, 300 mg) once daily taken as 1 capsule in the morning immediately before or within 1 hour after a meal, and matching placebo to asacol taken as 1 or 2 capsules TID as directed by the investigator for Week 1 to Week 6. Topical 5-ASA preparation was used as a rescue therapy.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg | Asacol | Total
Number analyzed (Participants) | 15 | 11 | 12 | 12 | 12 | 16 | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.0 (13.56) | 51.9 (9.59) | 53.4 (13.53) | 39.0 (11.17) | 42.0 (13.99) | 47.8 (13.34) | 46.1 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 2 | 2 | 5 | 8 | 24
  Male | 13 | 6 | 10 | 10 | 7 | 8 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 0 | 1 | 3
  White | 14 | 11 | 12 | 10 | 11 | 13 | 71
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AE) or Serious Adverse Events (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, associated with liver injury and impaired liver function defined as alanine aminotransferase >=3 x upper limit of normal (ULN), and total bilirubin >=2 x ULN or international normalized ratio >1.5.
Time Frame: Up to Week 6
Population: Intent-To-Treat (ITT) Population was defined as all participants who were randomized to treatment, who received at least one dose of study medication and who had at least one valid post dose assessment.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg | Asacol
Number analyzed (Participants) | 15 | 11 | 12 | 12 | 12 | 16
Participants
  Any AE | 10 | 7 | 9 | 6 | 5 | 12
  Any SAE | 1 | 2 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Clinical Chemistry Data Outside the Reference Range
Description: Normal reference range for clinical chemistry parameters include: alanine amino transferase (ALT) 0-41 international units per liter (IU/L); aspartate amino transferase (AST) 10 - 38 IU/L; alkaline phosphatase 40 - 129 IU/L; gamma glutamyl transferase (GGT) 10 - 66 IU/L; albumin 39 - 48 gram per liter (g/L); total protein 66 - 87 g/L; direct bilirubin 0 - 5.13 micromole per liter (µmol/L); total bilirubin 0 - 17.1 µmol/L; creatinine 61.88 - 106.08 µmol/L; uric acid 202.232 - 416.36 µmol/L; calcium 2.0958 - 2.42015 millimole per liter (mmol/L); cholesterol 2.8446 - 5.9478 mmol/L; chloride 98 - 106 mmol/L; glucose 2.2204 - 11.102 mmol/L; potassium 3.4 - 4.5 mmol/L; magnesium 0.6576 - 1.0686 mmol/L; sodium 0 - 2.26 mmol/L; urea/ blood urea nitrogen (BUN) 0 - 17.85 mmol/L. Number of participants with high and low values compared to the reference range is presented. Only those parameters for which at least one value outside the reference range was reported at any visit are summarized.
Time Frame: Screening (Day -7 to -1), Day 1, Week 1, 2, 3, 4 and 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg | Asacol
Number analyzed (Participants) | 15 | 11 | 12 | 12 | 12 | 16
Participants
  ALT, Week 6, high: number analyzed (Participants) | 13 | 7 | 8 | 10 | 9 | 12
  ALT, Week 6, high | 0 | 0 | 1 | 0 | 0 | 0
  Albumin, Screening, low: number analyzed (Participants) | 15 | 7 | 11 | 10 | 11 | 16
  Albumin, Screening, low | 0 | 0 | 1 | 0 | 0 | 1
  Albumin, Week 2, low: number analyzed (Participants) | 15 | 8 | 10 | 11 | 9 | 13
  Albumin, Week 2, low | 0 | 0 | 1 | 0 | 1 | 0
  Albumin, Week 4, low: number analyzed (Participants) | 15 | 5 | 11 | 11 | 9 | 13
  Albumin, Week 4, low | 0 | 0 | 1 | 0 | 1 | 1
  Albumin, Week 6, low: number analyzed (Participants) | 13 | 5 | 6 | 9 | 9 | 12
  Albumin, Week 6, low | 0 | 0 | 1 | 0 | 1 | 1
  Calcium, Week 2, high: number analyzed (Participants) | 15 | 10 | 11 | 11 | 9 | 13
  Calcium, Week 2, high | 1 | 0 | 0 | 0 | 0 | 0
  Calcium, Week 4, high: number analyzed (Participants) | 15 | 7 | 12 | 11 | 8 | 12
  Calcium, Week 4, high | 1 | 0 | 0 | 0 | 0 | 0
  Calcium, Week 6, high: number analyzed (Participants) | 13 | 7 | 7 | 9 | 8 | 12
  Calcium, Week 6, high | 1 | 0 | 0 | 0 | 0 | 0
  Glucose, Screening, high: number analyzed (Participants) | 14 | 9 | 11 | 10 | 12 | 15
  Glucose, Screening, high | 0 | 0 | 0 | 0 | 1 | 0
  Glucose, Week 2, high: number analyzed (Participants) | 15 | 10 | 12 | 11 | 9 | 14
  Glucose, Week 2, high | 0 | 0 | 1 | 0 | 1 | 0
  Magnesium, Week 2, high: number analyzed (Participants) | 15 | 9 | 12 | 11 | 9 | 13
  Magnesium, Week 2, high | 0 | 0 | 0 | 1 | 0 | 0
  Magnesium, Week 2, low: number analyzed (Participants) | 15 | 9 | 12 | 11 | 9 | 13
  Magnesium, Week 2, low | 0 | 0 | 0 | 0 | 0 | 1
  Potassium, Week 6, high: number analyzed (Participants) | 13 | 7 | 8 | 10 | 9 | 11
  Potassium, Week 6, high | 0 | 1 | 0 | 0 | 0 | 0
  Sodium, Screening, low: number analyzed (Participants) | 15 | 11 | 12 | 11 | 11 | 16
  Sodium, Screening, low | 0 | 0 | 1 | 0 | 0 | 0
  Total Bilirubin, Week 4, high: number analyzed (Participants) | 15 | 7 | 12 | 11 | 9 | 12
  Total Bilirubin, Week 4, high | 1 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Hematology Data Outside the Reference Range
Description: Normal reference range for clinical chemistry parameters include: basophils 0 - 0.2 giga cells (GI)/L; eosinophils 0 - 0.4 GI/L; lymphocytes 1 - 4.8 GI/L; monocyte 0 - 0.8 GI/L; total neutrophils (total absolute neutrophils count) 1.8 - 7.7 GI/L; platelet count 150 - 400 GI/L; red blood cell count 4.5 - 5.9 GI/L; white blood cell count 3.9 - 10.6 GI/L; hemoglobin 135 - 175 g/L; hematocrit 0.41 - 0.53 ratio; mean corpuscle hemoglobin concentration 310 - 370 g/L; mean corpuscle hemoglobin 26 - 34 picogram (PG); mean corpuscle volume 80 - 100 femtoliter (FL); reticulocytes 0.05 - 0.1 trillion cells (TI)/L. Number of participants with high and low values compared to the reference range is presented. Only those parameters for which at least one value outside the reference range was reported at any visit are summarized.
Time Frame: Screening (Day -7 to -1), Day 1, Week 1, 2, 3, 4 and 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg | Asacol
Number analyzed (Participants) | 15 | 11 | 12 | 12 | 12 | 16
Participants
  Lymphocytes, Screening, low: number analyzed (Participants) | 15 | 11 | 12 | 11 | 11 | 16
  Lymphocytes, Screening, low | 0 | 1 | 1 | 2 | 3 | 3
  Lymphocytes, Week 1, low: number analyzed (Participants) | 13 | 9 | 12 | 12 | 11 | 14
  Lymphocytes, Week 1, low | 0 | 1 | 3 | 2 | 2 | 3
  Lymphocytes, Week 2, low: number analyzed (Participants) | 15 | 9 | 12 | 11 | 10 | 14
  Lymphocytes, Week 2, low | 0 | 1 | 2 | 1 | 3 | 1
  Lymphocytes, Week 4, low: number analyzed (Participants) | 15 | 6 | 12 | 11 | 9 | 13
  Lymphocytes, Week 4, low | 1 | 1 | 3 | 1 | 4 | 1
  Lymphocytes, Week 6, low: number analyzed (Participants) | 13 | 7 | 8 | 10 | 9 | 13
  Lymphocytes, Week 6, low | 0 | 1 | 1 | 1 | 2 | 1
  Platelet count, Screening, high | 0 | 0 | 0 | 0 | 1 | 0
  Platelet count, Week 1, high: number analyzed (Participants) | 13 | 9 | 12 | 12 | 11 | 14
  Platelet count, Week 1, high | 0 | 0 | 0 | 0 | 1 | 0
  Platelet count, Week 2, high: number analyzed (Participants) | 15 | 10 | 12 | 11 | 10 | 14
  Platelet count, Week 2, high | 0 | 0 | 0 | 0 | 1 | 0
  Platelet count, Week 4, high: number analyzed (Participants) | 15 | 7 | 12 | 11 | 9 | 13
  Platelet count, Week 4, high | 0 | 0 | 0 | 0 | 1 | 0
  Platelet count, Week 6, high: number analyzed (Participants) | 13 | 7 | 8 | 10 | 9 | 13
  Platelet count, Week 6, high | 0 | 0 | 0 | 0 | 1 | 0
  Total ANC, Screening, low: number analyzed (Participants) | 15 | 11 | 11 | 11 | 11 | 16
  Total ANC, Screening, low | 1 | 0 | 0 | 0 | 0 | 0
  WBC, Screening, low | 1 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants of Abnormal Urinalysis Dipstick Results
Description: The urinalysis parameters included urine occult blood, urine general, glucose, ketones and protein by dipstick analysis. The assessments were done on screening, Week 2, Week 4 and Week 6.The number of participants with results of 0, 0.3, 1, 1+, 1.5, 10, 2+, 3+, 30, 4+, 5+, 55, not rated (NR), positive (pos) and trace is presented.
Time Frame: Screening (Day -7 to -1), Week 2, 4 and 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg | Asacol
Number analyzed (Participants) | 15 | 11 | 12 | 12 | 12 | 16
Participants
  Occult Blood, Screening, 0: number analyzed (Participants) | 14 | 11 | 12 | 12 | 11 | 15
  Occult Blood, Screening, 0 | 3 | 0 | 2 | 0 | 1 | 1
  Occult Blood, Screening, 1+: number analyzed (Participants) | 14 | 11 | 12 | 12 | 11 | 15
  Occult Blood, Screening, 1+ | 1 | 0 | 1 | 1 | 0 | 0
  Occult Blood, Screening, 2+: number analyzed (Participants) | 14 | 11 | 12 | 12 | 11 | 15
  Occult Blood, Screening, 2+ | 0 | 0 | 0 | 0 | 0 | 1
  Occult Blood, Screening, 5+: number analyzed (Participants) | 14 | 11 | 12 | 12 | 11 | 15
  Occult Blood, Screening, 5+ | 0 | 0 | 0 | 0 | 0 | 1
  Occult Blood, Screening, Pos: number analyzed (Participants) | 14 | 11 | 12 | 12 | 11 | 15
  Occult Blood, Screening, Pos | 0 | 0 | 0 | 0 | 2 | 1
  Occult Blood, Screening, Trace: number analyzed (Participants) | 14 | 11 | 12 | 12 | 11 | 15
  Occult Blood, Screening, Trace | 1 | 3 | 1 | 0 | 0 | 1
  Occult Blood, Week 2, 0: number analyzed (Participants) | 14 | 10 | 11 | 11 | 9 | 14
  Occult Blood, Week 2, 0 | 2 | 0 | 2 | 0 | 1 | 1
  Occult Blood, Week 2, 2+: number analyzed (Participants) | 14 | 10 | 11 | 11 | 9 | 14
  Occult Blood, Week 2, 2+ | 0 | 0 | 0 | 1 | 0 | 0
  Occult Blood, Week 2, 4+: number analyzed (Participants) | 14 | 10 | 11 | 11 | 9 | 14
  Occult Blood, Week 2, 4+ | 0 | 0 | 0 | 0 | 0 | 1
  Occult Blood, Week 2, Pos: number analyzed (Participants) | 14 | 10 | 11 | 11 | 9 | 14
  Occult Blood, Week 2, Pos | 0 | 0 | 1 | 0 | 0 | 0
  Occult Blood, Week 2, trace: number analyzed (Participants) | 14 | 10 | 11 | 11 | 9 | 14
  Occult Blood, Week 2, trace | 1 | 3 | 0 | 0 | 0 | 1
  Occult Blood, Week 4, 0: number analyzed (Participants) | 14 | 7 | 9 | 11 | 9 | 13
  Occult Blood, Week 4, 0 | 3 | 0 | 1 | 0 | 1 | 1
  Occult Blood, Week 4, 2+: number analyzed (Participants) | 14 | 7 | 9 | 11 | 9 | 13
  Occult Blood, Week 4, 2+ | 0 | 0 | 1 | 0 | 0 | 0
  Occult Blood, Week 4, 3+: number analyzed (Participants) | 14 | 7 | 9 | 11 | 9 | 13
  Occult Blood, Week 4, 3+ | 0 | 0 | 0 | 0 | 1 | 0
  Occult Blood, Week 4, trace: number analyzed (Participants) | 14 | 7 | 9 | 11 | 9 | 13
  Occult Blood, Week 4, trace | 1 | 0 | 1 | 0 | 1 | 1
  Occult Blood, Week 6, 0: number analyzed (Participants) | 13 | 7 | 7 | 10 | 9 | 13
  Occult Blood, Week 6, 0 | 2 | 0 | 1 | 0 | 1 | 1
  Occult Blood, Week 6, 10: number analyzed (Participants) | 13 | 7 | 7 | 10 | 9 | 13
  Occult Blood, Week 6, 10 | 0 | 0 | 0 | 0 | 1 | 0
  Occult Blood, Week 6, trace: number analyzed (Participants) | 13 | 7 | 7 | 10 | 9 | 13
  Occult Blood, Week 6, trace | 0 | 0 | 1 | 0 | 1 | 0
  General, Screening, NR: number analyzed (Participants) | 14 | 11 | 12 | 12 | 12 | 16
  General, Screening, NR | 0 | 1 | 0 | 0 | 0 | 1
  General, Screening, Pos: number analyzed (Participants) | 14 | 11 | 12 | 12 | 12 | 16
  General, Screening, Pos | 2 | 4 | 5 | 2 | 2 | 4
  General, Week 2, NR: number analyzed (Participants) | 14 | 10 | 11 | 11 | 9 | 14
  General, Week 2, NR | 0 | 0 | 1 | 1 | 0 | 0
  General, Week 2, Pos: number analyzed (Participants) | 14 | 10 | 11 | 11 | 9 | 14
  General, Week 2, Pos | 3 | 2 | 2 | 1 | 0 | 3
  General, Week 4, NR: number analyzed (Participants) | 14 | 7 | 10 | 11 | 9 | 13
  General, Week 4, NR | 0 | 0 | 0 | 1 | 1 | 0
  General, Week 4, Pos: number analyzed (Participants) | 14 | 7 | 10 | 11 | 9 | 13
  General, Week 4, Pos | 3 | 2 | 4 | 2 | 2 | 3
  General, Week 6, NR: number analyzed (Participants) | 13 | 7 | 7 | 10 | 9 | 13
  General, Week 6, NR | 0 | 0 | 0 | 1 | 0 | 0
  General, Week 6, Pos: number analyzed (Participants) | 13 | 7 | 7 | 10 | 9 | 13
  General, Week 6, Pos | 3 | 0 | 1 | 0 | 1 | 3
  Glucose, Screening, 0: number analyzed (Participants) | 14 | 11 | 12 | 12 | 11 | 15
  Glucose, Screening, 0 | 3 | 0 | 3 | 1 | 1 | 2
  Glucose, Screening, 55: number analyzed (Participants) | 14 | 11 | 12 | 12 | 11 | 15
  Glucose, Screening, 55 | 0 | 0 | 0 | 0 | 1 | 0
  Glucose, Screening, Pos: number analyzed (Participants) | 14 | 11 | 12 | 12 | 11 | 15
  Glucose, Screening, Pos | 1 | 0 | 0 | 0 | 0 | 0
  Glucose, Week 2, 0: number analyzed (Participants) | 14 | 10 | 11 | 11 | 9 | 14
  Glucose, Week 2, 0 | 2 | 0 | 2 | 1 | 1 | 2
  Glucose, Week 2, Pos: number analyzed (Participants) | 14 | 10 | 11 | 11 | 9 | 14
  Glucose, Week 2, Pos | 0 | 0 | 1 | 0 | 0 | 0
  Glucose, Week 4, 0: number analyzed (Participants) | 14 | 7 | 9 | 11 | 9 | 13
  Glucose, Week 4, 0 | 3 | 0 | 1 | 1 | 1 | 2
  Glucose, Week 6, 0: number analyzed (Participants) | 13 | 7 | 7 | 10 | 9 | 13
  Glucose, Week 6, 0 | 2 | 0 | 1 | 1 | 1 | 2
  Glucose, Week 6, Pos: number analyzed (Participants) | 13 | 7 | 7 | 10 | 9 | 13
  Glucose, Week 6, Pos | 0 | 0 | 1 | 0 | 0 | 0
  Ketones, Screening, 0: number analyzed (Participants) | 14 | 11 | 11 | 12 | 11 | 15
  Ketones, Screening, 0 | 1 | 0 | 1 | 1 | 0 | 0
  Ketones, Screening, 3+: number analyzed (Participants) | 14 | 11 | 11 | 12 | 11 | 15
  Ketones, Screening, 3+ | 0 | 0 | 0 | 1 | 0 | 0
  Ketones, Screening, Pos: number analyzed (Participants) | 14 | 11 | 11 | 12 | 11 | 15
  Ketones, Screening, Pos | 0 | 2 | 1 | 0 | 0 | 1
  Ketones, Screening, Trace: number analyzed (Participants) | 14 | 11 | 11 | 12 | 11 | 15
  Ketones, Screening, Trace | 0 | 0 | 0 | 1 | 1 | 0
  Ketones, Week 2, 0: number analyzed (Participants) | 14 | 10 | 10 | 11 | 9 | 14
  Ketones, Week 2, 0 | 0 | 0 | 0 | 1 | 0 | 0
  Ketones, Week 2, 1+: number analyzed (Participants) | 14 | 10 | 10 | 11 | 9 | 14
  Ketones, Week 2, 1+ | 0 | 0 | 0 | 0 | 0 | 1
  Ketones, Week 2, Pos: number analyzed (Participants) | 14 | 10 | 10 | 11 | 9 | 14
  Ketones, Week 2, Pos | 0 | 0 | 0 | 0 | 1 | 0
  Ketones, Week 2, Trace: number analyzed (Participants) | 14 | 10 | 10 | 11 | 9 | 14
  Ketones, Week 2, Trace | 0 | 0 | 1 | 0 | 0 | 0
  Ketones, Week 4, 0: number analyzed (Participants) | 14 | 7 | 9 | 11 | 9 | 13
  Ketones, Week 4, 0 | 1 | 0 | 0 | 1 | 0 | 0
  Ketones, Week 4, 1.5: number analyzed (Participants) | 14 | 7 | 9 | 11 | 9 | 13
  Ketones, Week 4, 1.5 | 0 | 0 | 0 | 0 | 0 | 1
  Ketones, Week 6, 0: number analyzed (Participants) | 13 | 7 | 6 | 10 | 9 | 13
  Ketones, Week 6, 0 | 0 | 0 | 0 | 1 | 0 | 0
  Ketones, Week 6, 1+: number analyzed (Participants) | 13 | 7 | 6 | 10 | 9 | 13
  Ketones, Week 6, 1+ | 0 | 0 | 0 | 0 | 0 | 1
  Ketones, Week 6, Trace: number analyzed (Participants) | 13 | 7 | 6 | 10 | 9 | 13
  Ketones, Week 6, Trace | 0 | 0 | 0 | 0 | 0 | 1
  Protein, Screening, 0: number analyzed (Participants) | 14 | 11 | 12 | 11 | 11 | 14
  Protein, Screening, 0 | 3 | 0 | 3 | 1 | 1 | 1
  Protein, Screening, 0.3: number analyzed (Participants) | 14 | 11 | 12 | 11 | 11 | 14
  Protein, Screening, 0.3 | 0 | 0 | 0 | 1 | 0 | 0
  Protein, Screening, Pos: number analyzed (Participants) | 14 | 11 | 12 | 11 | 11 | 14
  Protein, Screening, Pos | 0 | 1 | 2 | 0 | 0 | 1
  Protein, Screening, Trace: number analyzed (Participants) | 14 | 11 | 12 | 11 | 11 | 14
  Protein, Screening, Trace | 2 | 1 | 0 | 0 | 2 | 1
  Protein, Week 2, 0: number analyzed (Participants) | 14 | 10 | 11 | 11 | 9 | 13
  Protein, Week 2, 0 | 2 | 0 | 2 | 1 | 1 | 1
  Protein, Week 2, Pos: number analyzed (Participants) | 14 | 10 | 11 | 11 | 9 | 13
  Protein, Week 2, Pos | 1 | 0 | 1 | 0 | 0 | 0
  Protein, Week 2, Trace: number analyzed (Participants) | 14 | 10 | 11 | 11 | 9 | 13
  Protein, Week 2, Trace | 2 | 1 | 0 | 0 | 0 | 1
  Protein, Week 4, 0: number analyzed (Participants) | 14 | 7 | 9 | 11 | 9 | 13
  Protein, Week 4, 0 | 3 | 0 | 1 | 1 | 1 | 2
  Protein, Week 4, 2+: number analyzed (Participants) | 14 | 7 | 9 | 11 | 9 | 13
  Protein, Week 4, 2+ | 0 | 0 | 0 | 0 | 0 | 1
  Protein, Week 4, 30: number analyzed (Participants) | 14 | 7 | 9 | 11 | 9 | 13
  Protein, Week 4, 30 | 0 | 0 | 1 | 0 | 0 | 0
  Protein, Week 4, Pos: number analyzed (Participants) | 14 | 7 | 9 | 11 | 9 | 13
  Protein, Week 4, Pos | 1 | 1 | 3 | 1 | 0 | 0
  Protein, Week 4, Trace: number analyzed (Participants) | 14 | 7 | 9 | 11 | 9 | 13
  Protein, Week 4, Trace | 3 | 0 | 0 | 1 | 0 | 0
  Protein, Week 6, 0: number analyzed (Participants) | 13 | 7 | 7 | 10 | 9 | 13
  Protein, Week 6, 0 | 2 | 0 | 1 | 1 | 1 | 1
  Protein, Week 6, 1: number analyzed (Participants) | 13 | 7 | 7 | 10 | 9 | 13
  Protein, Week 6, 1 | 0 | 0 | 0 | 0 | 1 | 0
  Protein, Week 6, Pos: number analyzed (Participants) | 13 | 7 | 7 | 10 | 9 | 13
  Protein, Week 6, Pos | 3 | 0 | 0 | 0 | 0 | 0
  Protein, Week 6, Trace: number analyzed (Participants) | 13 | 7 | 7 | 10 | 9 | 13
  Protein, Week 6, Trace | 0 | 0 | 0 | 0 | 0 | 2

5. Primary Outcome: Number of Participants With Vital Sign Outside Range of Potential Clinical Importance (PCI)
Description: Vital signs assessment included systolic blood pressure (SBP), Diastolic blood pressure (DBP) and heart rate (HR). Criteria for vital sign values meeting PCI included: SBP < 85 and > 160 millimeter of mercury (mmHg); DBP < 45 and > 100 mmHg and HR < 40 and > 110 beats per minute (bpm). The assessments were done on screening, Week 2, Week 4 and Week 6. The participants with values higher and lower than the PCI range is presented. Only those parameters for which at least one value of PCI was reported at any visit are summarized.
Time Frame: Screening (Day -7 to -1), Week 2, 4 and 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg | Asacol
Number analyzed (Participants) | 15 | 11 | 12 | 12 | 12 | 16
Participants
  SBP, Screening, > PCI range | 0 | 1 | 2 | 1 | 0 | 0
  SBP, Week 2, > PCI range: number analyzed (Participants) | 15 | 10 | 12 | 11 | 9 | 14
  SBP, Week 2, > PCI range | 0 | 0 | 0 | 1 | 0 | 0
  SBP, Week 4, > PCI range: number analyzed (Participants) | 14 | 7 | 12 | 11 | 9 | 13
  SBP, Week 4, > PCI range | 0 | 1 | 0 | 1 | 0 | 0
  SBP, Week 6, > PCI range: number analyzed (Participants) | 13 | 7 | 8 | 10 | 9 | 13
  SBP, Week 6, > PCI range | 0 | 1 | 1 | 0 | 0 | 0
  DBP, Screening, > PCI range | 1 | 0 | 0 | 0 | 0 | 0
  DBP, Week 4, > PCI range: number analyzed (Participants) | 14 | 7 | 12 | 11 | 9 | 13
  DBP, Week 4, > PCI range | 0 | 1 | 0 | 0 | 0 | 0
  DBP, Week 6, > PCI range: number analyzed (Participants) | 13 | 7 | 8 | 10 | 9 | 13
  DBP, Week 6, > PCI range | 1 | 0 | 0 | 0 | 0 | 0
  HR, Week 6, > PCI range: number analyzed (Participants) | 13 | 7 | 8 | 10 | 9 | 13
  HR, Week 6, > PCI range | 1 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Abnormal Electrocardiography (ECG) Findings
Description: Single 12-lead ECGs were obtained at each timepoint during the study using an ECG machine that automatically calculated the HR and measured PR, QRS, QT, and QTc intervals. Criteria for ECG parameter values meeting PCI included absolute QTc interval >500 millisecond (msec); increase from Baseline QTc >60 msec; PR interval <110 and >220 msec; QRS interval <75 and >110 msec. Only those participants for whom at least one value of abnormal clinically significant or abnormal not clinically significant ECG findings were reported at any visit are summarized.
Time Frame: Screening (Day -7 to -1), Week 2, 4 and 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg | Asacol
Number analyzed (Participants) | 15 | 11 | 12 | 12 | 12 | 16
Participants
  Not significant, Screening: number analyzed (Participants) | 15 | 10 | 12 | 12 | 12 | 16
  Not significant, Screening | 2 | 3 | 2 | 2 | 2 | 2
  Not significant, Week 2: number analyzed (Participants) | 15 | 10 | 12 | 11 | 9 | 14
  Not significant, Week 2 | 1 | 1 | 2 | 2 | 2 | 2
  Not significant, Week 4: number analyzed (Participants) | 15 | 7 | 12 | 10 | 9 | 13
  Not significant, Week 4 | 4 | 2 | 4 | 2 | 1 | 3
  Not significant, Week 6: number analyzed (Participants) | 13 | 7 | 8 | 10 | 9 | 13
  Not significant, Week 6 | 2 | 2 | 2 | 1 | 1 | 5

7. Primary Outcome: Mean Treatment Effects on Basal Morning Cortisol and Adrenocorticotropic Hormone (ACTH) Stimulated Cortisol Levels at Week 4 in Comparison With Baseline
Description: Treatment effects was assessed using a low-dose ACTH stimulation test which was performed on Day 1 pre dose (Baseline) and at Week 4 visit. A blood sample for plasma cortisol was taken immediately, before and 30 minutes after an intravenous injection of 1 microgram (μg). tetracosactide acetate, a synthetic peptide displaying the same physiological properties as ACTH. The change from morning basal cortisol was calculated for Day 1 pre-dose (ACTH1) and Week 4 (ACTH2) using the equation: ACTH1 = Day 1 post ACTH - Day 1 pre ACTH; ACTH2 = Week 4 post ACTH - Week 4 pre ACTH. The change from morning basal cortisol between Week 4 and Day 1 (ACTH effect) was calculated as : ACTH effect = ACTH2 - ACTH1. The difference in morning basal cortisol between Week 4 and Day 1 (ACTH morning) was calculated as:- ACTH morning = Week 4 pre ACTH - Day 1 pre ACTH. Adrenocorticol function was classed as normal if the change from post ACTH to pre ACTH (using ACTH1 and ACTH2) was >= 200 nanomoles per liter.
Time Frame: Baseline (Day 1, pre dose) and Week 4
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Nanomoles per liter
Arm/Group | Placebo | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg | Asacol
Number analyzed (Participants) | 15 | 11 | 12 | 12 | 12 | 16
Nanomoles per liter
  ACTH 1 | 180.1 (68.48) | 105.2 (79.96) | 304.3 (76.56) | -4.9 (76.56) | 310.5 (76.56) | 312.8 (66.30)
  ACTH 2: number analyzed (Participants) | 11 | 6 | 9 | 10 | 9 | 12
  ACTH 2 | 243.1 (81.06) | 152.7 (110.47) | 167.6 (92.42) | 188.6 (88.12) | 307.8 (97.42) | 143.4 (81.06)
  ACTH effect: number analyzed (Participants) | 11 | 6 | 9 | 10 | 9 | 12
  ACTH effect | 96.1 (103.99) | -29.4 (141.71) | -181.8 (118.57) | 217.8 (113.05) | 22.6 (124.98) | -152.4 (103.99)
  ACTH morning: number analyzed (Participants) | 11 | 6 | 9 | 10 | 9 | 12
  ACTH morning | -48.8 (64.95) | -16.6 (88.51) | 116.5 (74.05) | -202.2 (70.60) | -44.1 (78.06) | 71.1 (64.95)
Statistical Analysis 1: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for ACTH 1; Test type: Superiority or Other; p = 0.4788, Mixed Models Analysis; Mean Difference (Net) = -75.0, 95% CI 2-sided [-284.8 to 134.9]
Statistical Analysis 2: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for ACTH 1; Test type: Superiority or Other; p = 0.2309, Mixed Models Analysis; Mean Difference (Net) = 124.1, 95% CI 2-sided [-80.6 to 328.9]
Statistical Analysis 3: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for ACTH 1; Test type: Superiority or Other; p = 0.0758, Mixed Models Analysis; Mean Difference (Net) = -185.1, 95% CI 2-sided [-389.8 to 19.7]
Statistical Analysis 4: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for ACTH 1; Test type: Superiority or Other; p = 0.2084, Mixed Models Analysis; Median Difference (Net) = 130.4, 95% CI 2-sided [-74.4 to 335.1]
Statistical Analysis 5: Comparison: Placebo vs Asacol; Placebo versus Asacol for ACTH 1; Test type: Superiority or Other; p = 0.1684, Mixed Models Analysis; Mean Difference (Net) = 132.6, 95% CI 2-sided [-57.4 to 322.6]
Statistical Analysis 6: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for ACTH 2; Test type: Superiority or Other; p = 0.5122, Mixed Models Analysis; Mean Difference (Net) = -90.4, 95% CI 2-sided [-364.7 to 184.0]
Statistical Analysis 7: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for ACTH 2; Test type: Superiority or Other; p = 0.5417, Mixed Models Analysis; Mean Difference (Net) = -75.5, 95% CI 2-sided [-321.7 to 170.7]
Statistical Analysis 8: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for ACTH 2; Test type: Superiority or Other; p = 0.6511, Mixed Models Analysis; Mean Difference (Net) = -54.4, 95% CI 2-sided [-294.2 to 185.3]
Statistical Analysis 9: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for ACTH 2; Test type: Superiority or Other; p = 0.6117, Mixed Models Analysis; Mean Difference (Net) = 64.7, 95% CI 2-sided [-189.1 to 318.5]
Statistical Analysis 10: Comparison: Placebo vs Asacol; Placebo versus Asacol for ACTH 2; Test type: Superiority or Other; p = 0.3882, Mixed Models Analysis; Mean Difference (Net) = -99.7, 95% CI 2-sided [-329.3 to 129.9]
Statistical Analysis 11: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for ACTH effect; Test type: Superiority or Other; p = 0.4781, Mixed Models Analysis; Mean Difference (Net) = -125.5, 95% CI 2-sided [-477.5 to 226.5]
Statistical Analysis 12: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for ACTH effect; Test type: Superiority or Other; p = 0.0834, Mixed Models Analysis; Mean Difference (Net) = -277.9, 95% CI 2-sided [-593.7 to 37.9]
Statistical Analysis 13: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for ACTH effect; Test type: Superiority or Other; p = 0.4313, Mixed Models Analysis; Mean Difference (Net) = 121.7, 95% CI 2-sided [-185.8 to 429.3]
Statistical Analysis 14: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for ACTH effect; Test type: Superiority or Other; p = 0.6528, Mixed Models Analysis; Mean Difference (Net) = -73.5, 95% CI 2-sided [-399.1 to 252.0]
Statistical Analysis 15: Comparison: Placebo vs Asacol; Placebo versus Asacol for ACTH effect; Test type: Superiority or Other; p = 0.0966, Mixed Models Analysis; Mean Difference (Net) = -248.5, 95% CI 2-sided [-542.9 to 46.0]
Statistical Analysis 16: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for ACTH morning; Test type: Superiority or Other; p = 0.7704, Mixed Models Analysis; Mean Difference (Net) = 32.2, 95% CI 2-sided [-187.6 to 252.0]
Statistical Analysis 17: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for ACTH morning; Test type: Superiority or Other; p = 0.0988, Mixed Models Analysis; Mean Difference (Net) = 165.3, 95% CI 2-sided [-32.0 to 362.5]
Statistical Analysis 18: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for ACTH morning; Test type: Superiority or Other; p = 0.1153, Mixed Models Analysis; Mean Difference (Net) = -153.4, 95% CI 2-sided [-345.5 to 38.7]
Statistical Analysis 19: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for ACTH morning; Test type: Superiority or Other; p = 0.9636, Mixed Models Analysis; Mean Difference (Net) = 4.7, 95% CI 2-sided [-198.7 to 208.0]
Statistical Analysis 20: Comparison: Placebo vs Asacol; Placebo versus Asacol for ACTH morning; Test type: Superiority or Other; p = 0.1972, Mixed Models Analysis; Mean Difference (Net) = 119.8, 95% CI 2-sided [-64.1 to 303.8]
Statistical Analysis 21: Comparison: GSK1399686 10 mg vs Asacol; Asacol versus GSK1399686 10 mg for ACTH 1; Test type: Superiority or Other; p = 0.0495, Mixed Models Analysis; Mean Difference (Net) = -207.6, 95% CI 2-sided [-414.6 to -0.5]
Statistical Analysis 22: Comparison: GSK1399686 30 mg vs Asacol; Asacol versus GSK1399686 30 mg for ACTH 1; Test type: Superiority or Other; p = 0.9333, Mixed Models Analysis; Mean Difference (Net) = -8.5, 95% CI 2-sided [-210.4 to 193.4]
Statistical Analysis 23: Comparison: GSK1399686 100 mg vs Asacol; Asacol versus GSK1399686 100 mg for ACTH 1; Test type: Superiority or Other; p = 0.0025, Mixed Models Analysis; Mean Difference (Net) = -317.7, 95% CI 2-sided [-519.6 to -115.8]
Statistical Analysis 24: Comparison: GSK1399686 300 mg vs Asacol; Asacol versus GSK1399686 300 mg for ACTH 1; Test type: Superiority or Other; p = 0.9823, Mixed Models Analysis; Mean Difference (Net) = -2.2, 95% CI 2-sided [-204.1 to 199.6]
Statistical Analysis 25: Comparison: GSK1399686 10 mg vs Asacol; Asacol versus GSK1399686 10 mg for ACTH 2; Test type: Superiority or Other; p = 0.9460, Mixed Models Analysis; Mean Difference (Net) = 9.3, 95% CI 2-sided [-265.0 to 283.7]
Statistical Analysis 26: Comparison: GSK1399686 30 mg vs Asacol; Asacol versus GSK1399686 30 mg for ACTH 2; Test type: Superiority or Other; p = 0.8445, Mixed Models Analysis; Mean Difference (Net) = 24.2, 95% CI 2-sided [-222.0 to 270.4]
Statistical Analysis 27: Comparison: GSK1399686 100 mg vs Asacol; Asacol versus GSK1399686 100 mg for ACTH 2; Test type: Superiority or Other; p = 0.7069, Mixed Models Analysis; Mean Difference (Net) = 45.3, 95% CI 2-sided [-194.5 to 285.0]
Statistical Analysis 28: Comparison: GSK1399686 300 mg vs Asacol; Asacol versus GSK1399686 300 mg for ACTH 2; Test type: Superiority or Other; p = 0.1998, Mixed Models Analysis; Mean Difference (Net) = 164.4, 95% CI 2-sided [-89.4 to 418.2]
Statistical Analysis 29: Comparison: GSK1399686 10 mg vs Asacol; Asacol versus GSK1399686 10 mg for ACTH effect; Test type: Superiority or Other; p = 0.4871, Mixed Models Analysis; Mean Difference (Net) = 123.0, 95% CI 2-sided [-229.0 to 474.9]
Statistical Analysis 30: Comparison: GSK1399686 30 mg vs Asacol; Asacol versus GSK1399686 30 mg for ACTH effect; Test type: Superiority or Other; p = 0.8527, Mixed Models Analysis; Mean Difference (Net) = -29.4, 95% CI 2-sided [-345.2 to 286.4]
Statistical Analysis 31: Comparison: GSK1399686 100 mg vs Asacol; Asacol versus GSK1399686 100 mg for ACTH effect; Test type: Superiority or Other; p = 0.0192, Mixed Models Analysis; Mean Difference (Net) = 370.2, 95% CI 2-sided [62.6 to 677.8]
Statistical Analysis 32: Comparison: GSK1399686 300 mg vs Asacol; Asacol versus GSK1399686 300 mg for ACTH effect; Test type: Superiority or Other; p = 0.2865, Mixed Models Analysis; Mean Difference (Net) = 174.9, 95% CI 2-sided [-150.6 to 500.5]
Statistical Analysis 33: Comparison: GSK1399686 10 mg vs Asacol; Asacol versus GSK1399686 10 mg for ACTH morning; Test type: Superiority or Other; p = 0.4279, Mixed Models Analysis; Mean Difference (Net) = -87.6, 95% CI 2-sided [-307.5 to 132.2]
Statistical Analysis 34: Comparison: GSK1399686 30 mg vs Asacol; Asacol versus GSK1399686 30 mg for ACTH morning; Test type: Superiority or Other; p = 0.6464, Mixed Models Analysis; Mean Difference (Net) = 45.4, 95% CI 2-sided [-151.8 to 242.7]
Statistical Analysis 35: Comparison: GSK1399686 100 mg vs Asacol; Asacol versus GSK1399686 100 mg for ACTH morning; Test type: Superiority or Other; p = 0.0061, Mixed Models Analysis; Mean Difference (Net) = -273.3, 95% CI 2-sided [-465.4 to -81.2]
Statistical Analysis 36: Comparison: GSK1399686 300 mg vs Asacol; Asacol versus GSK1399686 300 mg for ACTH morning; Test type: Superiority or Other; p = 0.2614, Mixed Models Analysis; Mean Difference (Net) = -115.2, 95% CI 2-sided [-318.5 to 88.1]

8. Primary Outcome: Mean Concentration of GSK1399686 in Colon Biopsy Obtained Within 24 h After the Last Dose
Description: The assessment was done on the samples collected from the sigmoid colon and from the rectum obtained within 24 hour after the last dose on Week 4 visit after endoscopic evaluation of respective area for determination of GSK1399686 concentration. Non-quantifiable (NQ) concentration values were imputed as 0.
Time Frame: Week 4
Population: Pharmacokinetic (PK) Population which was defined as the participants in the ITT Population for whom a PK sample was obtained and analysed. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram (ng)/mL
Arm/Group | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg
Number analyzed (Participants) | 11 | 12 | 12 | 12
Nanogram (ng)/mL
  Rectum: number analyzed (Participants) | 6 | 8 | 7 | 9
  Rectum | 0.0222 (0.05430) | 3.9594 (6.78264) | 4.6149 (8.77772) | 22.9187 (31.33636)
  Sigmoid: number analyzed (Participants) | 5 | 8 | 7 | 9
  Sigmoid | 0.0652 (0.09284) | 4.9721 (7.84369) | 7.0701 (12.08217) | 24.2401 (19.50441)

9. Secondary Outcome: Mean Simple Clinical Colitis Activity Index (SCCAI) Score
Description: SSCAI included composite score: bowel frequency during day on a scale of 0-3 defined as 0 was <= 3, 1= 4 to 6, 2= 7 to 9 and 3 was > 9, during night on a scale of 0-2 defined as 0= none, 1=1 to 3 and 2 was >=4, defecation urgency on a scale of 0-3 defined as 0=none, 1=hurry, 2=immediately and 3=incontinence, blood in stool on a scale of 0-3 defined as 0= none, 1= trace, 2= occasionally frank and 3= usually frank, general well being on a scale of 0-4 defined as 0=very well, 1= slightly below par, 2= poor, 3 = very poor and 4= terrible, extracolonic features (arthritis, pyoderma gangrenosum, erythema nodosum, uveitis) on a scale of 0-1 defined as 0= absent, 1= present. The SCCAI score was calculated as a sum of scores for each individual component of the SCCAI. Minimum score 0, maximum score 19. Higher score implied worsening of symptoms. Participants were given a diary to score each component of SCCAI each morning. Average SCCAI scores over last 3 days were used for each Week.
Time Frame: Up to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed. Analysis was done on OC data referred to data collected on the electronic case report form (eCRF) without any imputations added.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg | Asacol
Number analyzed (Participants) | 15 | 11 | 12 | 12 | 12 | 16
Score on scale
  Week 1: number analyzed (Participants) | 15 | 10 | 12 | 12 | 11 | 15
  Week 1 | 4.3 (0.58) | 4.1 (0.67) | 5.7 (0.67) | 4.8 (0.67) | 5.3 (0.68) | 4.5 (0.55)
  Week 2: number analyzed (Participants) | 15 | 10 | 12 | 11 | 9 | 15
  Week 2 | 4.3 (0.63) | 4.6 (0.73) | 5.2 (0.73) | 3.9 (0.75) | 5.0 (0.79) | 3.7 (0.60)
  Week 3: number analyzed (Participants) | 14 | 7 | 12 | 11 | 9 | 14
  Week 3 | 4.4 (0.66) | 4.5 (0.82) | 5.4 (0.76) | 4.0 (0.78) | 5.2 (0.83) | 3.9 (0.63)
  Week 4: number analyzed (Participants) | 14 | 7 | 10 | 11 | 9 | 13
  Week 4 | 3.4 (0.73) | 4.6 (0.89) | 4.6 (0.85) | 3.7 (0.87) | 4.5 (0.91) | 3.8 (0.70)
  Week 5: number analyzed (Participants) | 13 | 6 | 8 | 10 | 9 | 12
  Week 5 | 3.7 (0.79) | 5.0 (0.98) | 4.3 (0.95) | 3.9 (0.95) | 4.2 (0.98) | 3.2 (0.77)
  Week 6: number analyzed (Participants) | 13 | 6 | 8 | 9 | 9 | 12
  Week 6 | 3.9 (0.79) | 4.5 (1.01) | 4.4 (0.96) | 3.7 (0.95) | 4.5 (0.99) | 3.1 (0.77)
Statistical Analysis 1: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 1 SCCAI score; Test type: Superiority or Other; p = 0.7559, Repeated measures mixed model — Analysis was adjusted for baseline (Day -1) SCCAI score, Baseline (Screening) Endoscopy Score and Baseline (Screening) UCDAI Score; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-2.0 to 1.5]
Statistical Analysis 2: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 1 SCCAI score; Test type: Superiority or Other; p = 0.1238, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-0.4 to 3.2]
Statistical Analysis 3: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 1 SCCAI score; Test type: Superiority or Other; p = 0.6302, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.3 to 2.2]
Statistical Analysis 4: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 1 SCCAI score; Test type: Superiority or Other; p = 0.2777, Repeated measures mixed model; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-0.8 to 2.8]
Statistical Analysis 5: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 1 SCCAI score; Test type: Superiority or Other; p = 0.8069, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.4 to 1.8]
Statistical Analysis 6: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 2 SCCAI score; Test type: Superiority or Other; p = 0.7699, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.6 to 2.2]
Statistical Analysis 7: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 2 SCCAI score; Test type: Superiority or Other; p = 0.3869, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-1.1 to 2.8]
Statistical Analysis 8: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 2 SCCAI score; Test type: Superiority or Other; p = 0.6695, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.4 to 1.5]
Statistical Analysis 9: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 2 SCCAI score; Test type: Superiority or Other; p = 0.5152, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-1.4 to 2.7]
Statistical Analysis 10: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 2 SCCAI score; Test type: Superiority or Other; p = 0.4507, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-2.4 to 1.1]
Statistical Analysis 11: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 3 SCCAI score; Test type: Superiority or Other; p = 0.8707, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.9 to 2.3]
Statistical Analysis 12: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 3 SCCAI score; Test type: Superiority or Other; p = 0.2915, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-0.9 to 3.1]
Statistical Analysis 13: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 3 SCCAI score; Test type: Superiority or Other; p = 0.7251, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.4 to 1.7]
Statistical Analysis 14: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 3 SCCAI score; Test type: Superiority or Other; p = 0.4556, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-1.3 to 2.9]
Statistical Analysis 15: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 3 SCCAI score; Test type: Superiority or Other; p = 0.6620, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.3 to 1.4]
Statistical Analysis 16: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 4 SCCAI score; Test type: Superiority or Other; p = 0.2844, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-1.1 to 3.5]
Statistical Analysis 17: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 4 SCCAI score; Test type: Superiority or Other; p = 0.2799, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-1.0 to 3.5]
Statistical Analysis 18: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 4 SCCAI score; Test type: Superiority or Other; p = 0.7655, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.9 to 2.6]
Statistical Analysis 19: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 4 SCCAI score; Test type: Superiority or Other; p = 0.3332, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-1.2 to 3.5]
Statistical Analysis 20: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 4 SCCAI score; Test type: Superiority or Other; p = 0.6985, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.6 to 2.4]
Statistical Analysis 21: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 5 SCCAI score; Test type: Superiority or Other; p = 0.3256, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-1.3 to 3.7]
Statistical Analysis 22: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 5 SCCAI score; Test type: Superiority or Other; p = 0.6500, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-1.9 to 3.0]
Statistical Analysis 23: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 5 SCCAI score; Test type: Superiority or Other; p = 0.8758, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-2.3 to 2.7]
Statistical Analysis 24: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 5 SCCAI score; Test type: Superiority or Other; p = 0.7298, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-2.1 to 3.0]
Statistical Analysis 25: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 5 SCCAI score; Test type: Superiority or Other; p = 0.5963, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.8 to 1.6]
Statistical Analysis 26: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 6 SCCAI score; Test type: Superiority or Other; p = 0.6498, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-2.0 to 3.1]
Statistical Analysis 27: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 6 SCCAI score; Test type: Superiority or Other; p = 0.7061, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-2.0 to 3.0]
Statistical Analysis 28: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 6 SCCAI score; Test type: Superiority or Other; p = 0.8549, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.7 to 2.3]
Statistical Analysis 29: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 6 SCCAI score; Test type: Superiority or Other; p = 0.6533, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-2.0 to 3.1]
Statistical Analysis 30: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 6 SCCAI score; Test type: Superiority or Other; p = 0.4378, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-3.1 to 1.4]
Statistical Analysis 31: Comparison: GSK1399686 10 mg vs Asacol; Asacol versus GSK1399686 10 mg for Week 1 SCCAI score; Test type: Superiority or Other; p = 0.5917, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-2.2 to 1.3]
Statistical Analysis 32: Comparison: GSK1399686 30 mg vs Asacol; Asacol versus GSK1399686 30 mg for Week 1 SCCAI score; Test type: Superiority or Other; p = 0.1764, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-0.5 to 2.9]
Statistical Analysis 33: Comparison: GSK1399686 100 mg vs Asacol; Asacol versus GSK1399686 100 mg for Week 1 SCCAI score; Test type: Superiority or Other; p = 0.7914, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.5 to 2.0]
Statistical Analysis 34: Comparison: GSK1399686 300 mg vs Asacol; Asacol versus GSK1399686 300 mg for Week 1 SCCAI score; Test type: Superiority or Other; p = 0.3578, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-0.9 to 2.5]
Statistical Analysis 35: Comparison: GSK1399686 10 mg vs Asacol; Asacol versus GSK1399686 10 mg for Week 2 SCCAI score; Test type: Superiority or Other; p = 0.3247, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-1.0 to 2.9]
Statistical Analysis 36: Comparison: GSK1399686 30 mg vs Asacol; Asacol versus GSK1399686 30 mg for Week 2 SCCAI score; Test type: Superiority or Other; p = 0.1153, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-0.4 to 3.4]
Statistical Analysis 37: Comparison: GSK1399686 100 mg vs Asacol; Asacol versus GSK1399686 100 mg for Week 2 SCCAI score; Test type: Superiority or Other; p = 0.7995, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.7 to 2.2]
Statistical Analysis 38: Comparison: GSK1399686 300 mg vs Asacol; Asacol versus GSK1399686 300 mg for Week 2 SCCAI score; Test type: Superiority or Other; p = 0.1786, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-0.6 to 3.3]
Statistical Analysis 39: Comparison: GSK1399686 10 mg vs Asacol; Asacol versus GSK1399686 10 mg for Week 3 SCCAI score; Test type: Superiority or Other; p = 0.5824, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-1.5 to 2.7]
Statistical Analysis 40: Comparison: GSK1399686 30 mg vs Asacol; Asacol versus GSK1399686 30 mg for Week 3 SCCAI score; Test type: Superiority or Other; p = 0.1392, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-0.5 to 3.5]
Statistical Analysis 41: Comparison: GSK1399686 100 mg vs Asacol; Asacol versus GSK1399686 100 mg for Week 3 SCCAI score; Test type: Superiority or Other; p = 0.9665, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-2.0 to 2.1]
Statistical Analysis 42: Comparison: GSK1399686 300 mg vs Asacol; Asacol versus GSK1399686 300 mg for Week 3 SCCAI score; Test type: Superiority or Other; p = 0.2455, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-0.9 to 3.3]
Statistical Analysis 43: Comparison: GSK1399686 10 mg vs Asacol; Asacol versus GSK1399686 10 mg for Week 4 SCCAI score; Test type: Superiority or Other; p = 0.4644, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-1.4 to 3.1]
Statistical Analysis 44: Comparison: GSK1399686 30 mg vs Asacol; Asacol versus GSK1399686 30 mg for Week 4 SCCAI score; Test type: Superiority or Other; p = 0.4567, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-1.4 to 3.0]
Statistical Analysis 45: Comparison: GSK1399686 100 mg vs Asacol; Asacol versus GSK1399686 100 mg for Week 4 SCCAI score; Test type: Superiority or Other; p = 0.9594, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-2.3 to 2.2]
Statistical Analysis 46: Comparison: GSK1399686 300 mg vs Asacol; Asacol versus GSK1399686 300 mg for Week 4 SCCAI score; Test type: Superiority or Other; p = 0.5122, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-1.5 to 3.0]
Statistical Analysis 47: Comparison: GSK1399686 10 mg vs Asacol; Asacol versus GSK1399686 10 mg for Week 5 SCCAI score; Test type: Superiority or Other; p = 0.1493, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-0.7 to 4.3]
Statistical Analysis 48: Comparison: GSK1399686 30 mg vs Asacol; Asacol versus GSK1399686 30 mg for Week 5 SCCAI score; Test type: Superiority or Other; p = 0.3478, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-1.3 to 3.6]
Statistical Analysis 49: Comparison: GSK1399686 100 mg vs Asacol; Asacol versus GSK1399686 100 mg for Week 5 SCCAI score; Test type: Superiority or Other; p = 0.5238, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-1.7 to 3.2]
Statistical Analysis 50: Comparison: GSK1399686 300 mg vs Asacol; Asacol versus GSK1399686 300 mg for Week 5 SCCAI score; Test type: Superiority or Other; p = 0.4091, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-1.4 to 3.5]
Statistical Analysis 51: Comparison: GSK1399686 10 mg vs Asacol; Asacol versus GSK1399686 10 mg for Week 6 SCCAI score; Test type: Superiority or Other; p = 0.2604, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-1.1 to 4.0]
Statistical Analysis 52: Comparison: GSK1399686 30 mg vs Asacol; Asacol versus GSK1399686 30 mg for Week 6 SCCAI score; Test type: Superiority or Other; p = 0.2809, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-1.1 to 3.8]
Statistical Analysis 53: Comparison: GSK1399686 100 mg vs Asacol; Asacol versus GSK1399686 100 mg for Week 6 SCCAI score; Test type: Superiority or Other; p = 0.6038, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-1.8 to 3.1]
Statistical Analysis 54: Comparison: GSK1399686 300 mg vs Asacol; Asacol versus GSK1399686 300 mg for Week 6 SCCAI score; Test type: Superiority or Other; p = 0.2511, Repeated measures mixed model — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-1.1 to 3.9]

10. Secondary Outcome: Number of Participants With Clinical Response and Clinical Remission at Week 4 and Week 6
Description: Participants were defined as clinical responders if the average change from baseline total SCCAI score was <-2. (i.e. the post dose total SCCAI score was decreased by >2 points compared to the baseline total SCCAI score). Baseline was defined as the value on Day -1. The change from baseline total SCCAI score was derived by subtracting the baseline value (Day -1) from the individual post-dose values. Participants were defined as in clinical remission if the post dose total SCCAI score was <3 and baseline SCCAI score was not <3 (i.e . =>3).
Time Frame: Week 4 and Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed. Analysis was done on OC data referred to data collected on the eCRF without any imputations added.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg | Asacol
Number analyzed (Participants) | 15 | 11 | 12 | 12 | 12 | 16
Participants
  Clinical Response, Week 4: number analyzed (Participants) | 14 | 7 | 10 | 11 | 9 | 13
  Clinical Response, Week 4 | 6 | 2 | 3 | 3 | 2 | 6
  Clinical Response, Week 6: number analyzed (Participants) | 13 | 6 | 8 | 9 | 9 | 12
  Clinical Response, Week 6 | 7 | 1 | 3 | 2 | 3 | 5
  Clinical Remission, Week 4: number analyzed (Participants) | 14 | 7 | 10 | 11 | 9 | 13
  Clinical Remission, Week 4 | 4 | 2 | 1 | 4 | 2 | 4
  Clinical Remission, Week 6: number analyzed (Participants) | 13 | 6 | 8 | 9 | 9 | 12
  Clinical Remission, Week 6 | 3 | 2 | 2 | 2 | 3 | 7

11. Secondary Outcome: Median Time to Clinical Response and Clinical Remission
Description: Time to clinical response was defined as the number of days between first dose of study medication and first day of at least 3 consecutive days with SCCAI score decreased for >2 points in comparison with baseline (Day -1 value). Time to clinical remission was defined as the number of days between the first dose of study medication and the first day of at least 3 consecutive days with SCCAI score < 3. Time to clinical response and remission was derived using daily diary data. Participants who did not meet the criteria for clinical response or clinical remission were censored at their last day on study medication.
Time Frame: Up to Week 6
Population: ITT Population. Data is presented for the participants available at the time of assessment. Analysis was done on OC data referred to data collected on the eCRF without any imputations added.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg | Asacol
Number analyzed (Participants) | 13 | 8 | 8 | 8 | 9 | 13
Days
  Clinical response | 18.0 [2 to 45] | 16.5 [2 to 45] | 26.0 [8 to 44] | 27.5 [3 to 44] | 13.0 [2 to 45] | 22.0 [1 to 44]
  Clinical remission | 41.0 [6 to 46] | 16.5 [4 to 45] | 35.0 [21 to 44] | 20.5 [3 to 43] | 31.0 [2 to 45] | 23.0 [2 to 43]

12. Secondary Outcome: Mean Fecal Calprotectin Levels Over Time
Description: Fecal calprotectin, a non-invasive surrogate marker of inflammation in the small intestine, and levels of which was associated with mucosal healing. Calprotectin is a calcium and zinc-binding protein found in neutrophils, monocytes and macrophages. Calprotectin is produced in significant amounts by inflammatory cells. Fecal levels of this protein has been demonstrated to correlate with colorectal and intestinal inflammation. Calprotectin plays a regulatory role in the inflammatory process and used as a diagnostic biomarker. It was assessed from Week 1 to Week 6.
Time Frame: Up to Week 6
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/g
Arm/Group | Placebo | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg | Asacol
Number analyzed (Participants) | 15 | 11 | 12 | 12 | 12 | 16
μg/g
  Week 1: number analyzed (Participants) | 15 | 10 | 12 | 12 | 11 | 15
  Week 1 | 1006.0 (131.15) | 553.6 (161.17) | 620.4 (380.26) | 453.5 (522.03) | 1173.2 (290.79) | 464.4 (238.45)
  Week 2: number analyzed (Participants) | 14 | 10 | 12 | 11 | 10 | 13
  Week 2 | 729.6 (279.89) | 514.0 (274.43) | 438.8 (321.40) | 303.6 (397.20) | 580.7 (259.64) | 419.3 (265.56)
  Week 3: number analyzed (Participants) | 13 | 6 | 9 | 10 | 9 | 13
  Week 3 | 829.9 (312.94) | 529.7 (305.31) | 525.4 (3600.04) | 404.5 (428.16) | 700.3 (279.46) | 289.2 (220.34)
  Week 4: number analyzed (Participants) | 14 | 6 | 10 | 10 | 9 | 13
  Week 4 | 651.3 (169.58) | 492.2 (644.48) | 431.3 (717.39) | 347.9 (842.92) | 908.9 (386.93) | 376.8 (329.51)
  Week 5: number analyzed (Participants) | 12 | 5 | 8 | 10 | 9 | 12
  Week 5 | 617.5 (156.54) | 246.1 (229.54) | 690.1 (1119.97) | 289.2 (524.84) | 347.7 (443.63) | 211.8 (637.18)
  Week 6: number analyzed (Participants) | 9 | 4 | 6 | 8 | 7 | 11
  Week 6 | 728.6 (214.08) | 276.2 (587.18) | 353.7 (960.48) | 142.9 (496.46) | 528.9 (184.78) | 347.4 (408.74)
Statistical Analysis 1: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 1 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.75, 95% CI 2-sided [0.24 to 2.39]
Statistical Analysis 2: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 1 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.64, 95% CI 2-sided [0.21 to 1.92]
Statistical Analysis 3: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 1 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.80, 95% CI 2-sided [0.26 to 2.48]
Statistical Analysis 4: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 1 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.85, 95% CI 2-sided [0.27 to 2.68]
Statistical Analysis 5: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 1 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.64, 95% CI 2-sided [0.23 to 1.81]
Statistical Analysis 6: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 2 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.85, 95% CI 2-sided [0.26 to 2.73]
Statistical Analysis 7: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 2 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.55, 95% CI 2-sided [0.18 to 1.68]
Statistical Analysis 8: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 2 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.67, 95% CI 2-sided [0.21 to 2.18]
Statistical Analysis 9: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 2 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.62, 95% CI 2-sided [0.19 to 2.03]
Statistical Analysis 10: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 2 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.64, 95% CI 2-sided [0.22 to 1.90]
Statistical Analysis 11: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 3 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 1.07, 95% CI 2-sided [0.28 to 4.09]
Statistical Analysis 12: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 3 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.74, 95% CI 2-sided [0.23 to 2.43]
Statistical Analysis 13: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 3 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.62, 95% CI 2-sided [0.18 to 2.08]
Statistical Analysis 14: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 3 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.60, 95% CI 2-sided [0.17 to 2.08]
Statistical Analysis 15: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 3 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.44, 95% CI 2-sided [0.15 to 1.32]
Statistical Analysis 16: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 4 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 1.29, 95% CI 2-sided [0.33 to 5.04]
Statistical Analysis 17: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 4 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.64, 95% CI 2-sided [0.20 to 2.02]
Statistical Analysis 18: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 4 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.96, 95% CI 2-sided [0.29 to 3.23]
Statistical Analysis 19: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 4 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 1.36, 95% CI 2-sided [0.39 to 4.72]
Statistical Analysis 20: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 4 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.82, 95% CI 2-sided [0.28 to 2.42]
Statistical Analysis 21: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 5 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.61, 95% CI 2-sided [0.14 to 2.66]
Statistical Analysis 22: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 5 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 1.25, 95% CI 2-sided [0.35 to 4.38]
Statistical Analysis 23: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 5 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.71, 95% CI 2-sided [0.20 to 2.47]
Statistical Analysis 24: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 5 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.41, 95% CI 2-sided [0.11 to 1.46]
Statistical Analysis 25: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 5 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.47, 95% CI 2-sided [0.15 to 1.48]
Statistical Analysis 26: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 6 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.66, 95% CI 2-sided [0.13 to 3.39]
Statistical Analysis 27: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 6 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.44, 95% CI 2-sided [0.11 to 1.84]
Statistical Analysis 28: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 6 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.37, 95% CI 2-sided [0.09 to 1.48]
Statistical Analysis 29: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 6 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.76, 95% CI 2-sided [0.19 to 2.99]
Statistical Analysis 30: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 6 fecal calprotectin levels; Test type: Superiority or Other; Ratio = 0.72, 95% CI 2-sided [0.21 to 2.49]

13. Secondary Outcome: Mean Fecal Lactoferrin Levels Over Time
Description: Fecal lactoferrin, a non-invasive surrogate marker of inflammation in the small intestine, and levels of which was associated with mucosal healing. Lactoferrin is an iron binding glycoprotein that is the major component of the secondary granules of polymorphonuclear neutrophils (but not monocytes and lymphocytes). Lactoferrin is produced in significant amounts by inflammatory cells. Fecal levels of this protein has been demonstrated to correlate with colorectal and intestinal inflammation. Lactoferrin plays an important role in the innate immunity as a bactericidal and used as a diagnostic biomarker. It was assessed from Week 1 to Week 6.
Time Frame: Up to Week 6
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/L
Arm/Group | Placebo | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg | Asacol
Number analyzed (Participants) | 15 | 11 | 12 | 12 | 12 | 16
µg/L
  Week 1: number analyzed (Participants) | 15 | 10 | 12 | 12 | 11 | 15
  Week 1 | 158.2 (300.88) | 166.1 (192.15) | 269.8 (664.28) | 163.0 (215.09) | 231.2 (201.16) | 175.3 (190.41)
  Week 2: number analyzed (Participants) | 14 | 10 | 12 | 11 | 10 | 13
  Week 2 | 194.7 (309.89) | 133.2 (259.95) | 148.7 (294.15) | 66.9 (408.38) | 150.2 (323.83) | 126.7 (368.30)
  Week 3: number analyzed (Participants) | 13 | 6 | 9 | 10 | 9 | 13
  Week 3 | 170.0 (303.14) | 76.5 (472.44) | 167.6 (440.45) | 105.8 (490.42) | 241.7 (269.59) | 52.9 (231.47)
  Week 4: number analyzed (Participants) | 14 | 6 | 9 | 10 | 9 | 13
  Week 4 | 166.0 (201.21) | 44.0 (104.68) | 126.4 (641.19) | 78.9 (538.99) | 177.5 (485.01) | 92.9 (313.55)
  Week 5: number analyzed (Participants) | 12 | 5 | 8 | 10 | 9 | 12
  Week 5 | 138.7 (244.59) | 145.8 (420.34) | 221.8 (184.47) | 47.1 (136.45) | 144.2 (276.04) | 102.0 (344.29)
  Week 6: number analyzed (Participants) | 9 | 4 | 5 | 8 | 7 | 11
  Week 6 | 89.1 (524.87) | 116.9 (548.47) | 207.9 (169.80) | 42.8 (261.57) | 127.3 (187.33) | 80.8 (186.07)
Statistical Analysis 1: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 1 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 1.19, 95% CI 2-sided [0.42 to 3.38]
Statistical Analysis 2: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 1 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 1.35, 95% CI 2-sided [0.50 to 3.65]
Statistical Analysis 3: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 1 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 1.25, 95% CI 2-sided [0.45 to 3.47]
Statistical Analysis 4: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 1 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 1.26, 95% CI 2-sided [0.44 to 3.59]
Statistical Analysis 5: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 1 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 1.28, 95% CI 2-sided [0.50 to 3.28]
Statistical Analysis 6: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 2 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.76, 95% CI 2-sided [0.26 to 2.19]
Statistical Analysis 7: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 2 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.59, 95% CI 2-sided [0.22 to 1.63]
Statistical Analysis 8: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 2 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.35, 95% CI 2-sided [0.12 to 1.00]
Statistical Analysis 9: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 2 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.93, 95% CI 2-sided [0.31 to 2.77]
Statistical Analysis 10: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 2 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.70, 95% CI 2-sided [0.26 to 1.87]
Statistical Analysis 11: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 3 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.53, 95% CI 2-sided [0.15 to 1.84]
Statistical Analysis 12: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 3 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.96, 95% CI 2-sided [0.32 to 2.87]
Statistical Analysis 13: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 3 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.52, 95% CI 2-sided [0.17 to 1.56]
Statistical Analysis 14: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 3 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 1.42, 95% CI 2-sided [0.45 to 4.46]
Statistical Analysis 15: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 3 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.37, 95% CI 2-sided [0.14 to 1.01]
Statistical Analysis 16: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 4 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.33, 95% CI 2-sided [0.10 to 1.15]
Statistical Analysis 17: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 4 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.68, 95% CI 2-sided [0.23 to 2.03]
Statistical Analysis 18: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 4 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.56, 95% CI 2-sided [0.19 to 1.68]
Statistical Analysis 19: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 4 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 1.19, 95% CI 2-sided [0.38 to 3.70]
Statistical Analysis 20: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 4 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.71, 95% CI 2-sided [0.26 to 1.89]
Statistical Analysis 21: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 5 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 1.05, 95% CI 2-sided [0.27 to 4.07]
Statistical Analysis 22: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 5 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 1.48, 95% CI 2-sided [0.46 to 4.73]
Statistical Analysis 23: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 5 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.33, 95% CI 2-sided [0.11 to 1.02]
Statistical Analysis 24: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 5 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 1.16, 95% CI 2-sided [0.36 to 3.73]
Statistical Analysis 25: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 5 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.82, 95% CI 2-sided [0.29 to 2.33]
Statistical Analysis 26: Comparison: Placebo vs GSK1399686 10 mg; Placebo versus GSK1399686 10 mg for Week 6 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 1.44, 95% CI 2-sided [0.31 to 6.59]
Statistical Analysis 27: Comparison: Placebo vs GSK1399686 30 mg; Placebo versus GSK1399686 30 mg for Week 6 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 2.21, 95% CI 2-sided [0.54 to 9.04]
Statistical Analysis 28: Comparison: Placebo vs GSK1399686 100 mg; Placebo versus GSK1399686 100 mg for Week 6 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.41, 95% CI 2-sided [0.11 to 1.48]
Statistical Analysis 29: Comparison: Placebo vs GSK1399686 300 mg; Placebo versus GSK1399686 300 mg for Week 6 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 1.64, 95% CI 2-sided [0.46 to 5.91]
Statistical Analysis 30: Comparison: Placebo vs Asacol; Placebo versus Asacol for Week 6 fecal lactoferrin levels; Test type: Superiority or Other; Ratio = 0.84, 95% CI 2-sided [0.27 to 2.62]

14. Secondary Outcome: Mean Maximum Observed Concentration (Cmax) on Day 1 and Day 28 Derived From Observed Plasma Concentrations of GSK1399686 After Repeated Oral Dosing
Description: Cmax was derived on Day 1 and Day 28 from observed plasma concentrations of GSK1399686 after repeated oral dosing. Blood samples were collected on Day 1 (1 hour, 2 hour, 3 hour post dose) and Day 28 (Week 4 at pre dose, 1 hour, 2 hour, 3 hour and 4 hour morning post dose).
Time Frame: Day 1 (1 hour, 2 hour, 3 hour post dose) and Day 28 (Week 4 at pre dose, 1 hour, 2 hour, 3 hour and 4 hour morning post dose)
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram (ng)/mL
Arm/Group | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg
Number analyzed (Participants) | 11 | 12 | 12 | 12
Nanogram (ng)/mL
  Day 1: number analyzed (Participants) | 10 | 10 | 12 | 10
  Day 1 | 0.1326 (189.4) | 0.3854 (154.1) | 1.1309 (238.1) | 1.6866 (602.1)
  Day 28 (Week 4): number analyzed (Participants) | 7 | 10 | 11 | 9
  Day 28 (Week 4) | 0.1627 (155.5) | 0.1956 (485.5) | 0.6482 (306.2) | 5.5953 (107.6)

15. Secondary Outcome: Pre-dose Trough Concentration at the End of the Dosing Interval (Cτ) on Day 28 Derived From Observed Plasma Concentrations of GSK1399686 After Repeated Oral Dosing
Description: Cτ was derived on Day 28 from observed plasma concentrations of GSK1399686 after repeated oral dosing. Blood samples were collected on Day 28 (Week 4 at pre dose, 1 hour, 2 hour, 3 hour and 4 hour morning post dose).
Time Frame: Day 28 (Week 4 at pre dose, 1 hour, 2 hour, 3 hour and 4 hour morning post dose)
Population: PK Population. Data is presented for the participants available at the time of assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg
Number analyzed (Participants) | 7 | 9 | 11 | 9
ng/mL | 0.0500 (0.0) | 0.1294 (178.3) | 0.4930 (218.0) | 1.4066 (85.7)

16. Secondary Outcome: Plasma Clearance Estimated Based on Population Pharmacokinetic Analysis of Healthy Volunteers (Historical Data) and Patient Data
Description: Clearance derived from plasma concentration-time data was planned to be combined with data from healthy volunteers from Phase I study to characterize the population pharmacokinetics of GSK1399686. However data for this outcome measure was not collected.
Time Frame: Day 1 (1 hour, 2 hour, 3 hour post dose), Week 1 (anytime relative to the last dose), Week 2 (anytime relative to the last dose) and Day 28 (Week 4 at pre dose, 1 hour, 2 hour, 3 hour and 4 hour morning post dose)
Population: PK Population.
Groups:
- GSK1399686 10mg: Participants were administered oral dose of GSK1399686 10 mg QD in the morning for week 1 to week 4. Blinding was maintained by administration of matching placebo to asacol TID for week 1 to week 6 and matching placebo to GSK1399686 10 mg QD in the morning for week 5 to week 6. Topical 5-ASA preparation was used as a rescue therapy.
- GSK1399686 30mg: Participants were administered oral dose of GSK1399686 30 mg QD in the morning for week 1 to week 4. Blinding was maintained by administration of matching placebo to asacol TID for week 1 to week 6 and matching placebo to GSK1399686 30 mg QD in the morning for week 5 to week 6. Topical 5-ASA preparation was used as a rescue therapy.
- GSK1399686 100mg: Participants were administered oral dose of GSK1399686 100 mg QD in the morning for week 1 to week 4. Blinding was maintained by administration of matching placebo to asacol TID for week 1 to week 6 and matching placebo to GSK1399686 100 mg QD in the morning for week 5 to week 6. Topical 5-ASA preparation was used as a rescue therapy.
- GSK1399686 300mg: Participants were administered oral dose of GSK1399686 300 mg QD in the morning for week 1 to week 4. Blinding was maintained by administration of matching placebo to asacol TID for week 1 to week 6 and matching placebo to GSK1399686 300 mg QD in the morning for week 5 to week 6. Topical 5-ASA preparation was used as a rescue therapy.
Arm/Group | GSK1399686 10mg | GSK1399686 30mg | GSK1399686 100mg | GSK1399686 300mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Volume of Distribution Estimated Based on Population Pharmacokinetic Analysis of Healthy Volunteers (Historical Data) and Patient Data
Description: Volume of distribution derived from concentration-time data was planned to be combined with data from healthy volunteers from Phase I study to characterize the population pharmacokinetics of GSK1399686. However data for this outcome measure was not collected.
Time Frame: as for outcome 16
Population: PK Population.
Arm/Group | GSK1399686 10mg | GSK1399686 30mg | GSK1399686 100mg | GSK1399686 300mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AE's and SAE's were collected from from Screening (Day -7 to -1) to Week 6 (up to 45 days).
Description: ITT Population was used.
Arm/Group | Placebo | GSK1399686 10 mg | GSK1399686 30 mg | GSK1399686 100 mg | GSK1399686 300 mg | Asacol
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/11 | 0/12 | 0/12 | 0/12 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/15 | 2/11 | 0/12 | 0/12 | 0/12 | 1/16
Other Adverse Events (participants affected / at risk) | 10/15 | 6/11 | 9/12 | 6/12 | 5/12 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | GSK1399686 10 mg (N=11) | GSK1399686 30 mg (N=12) | GSK1399686 100 mg (N=12) | GSK1399686 300 mg (N=12) | Asacol (N=16)
Colitis ulcerative (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | GSK1399686 10 mg (N=11) | GSK1399686 30 mg (N=12) | GSK1399686 100 mg (N=12) | GSK1399686 300 mg (N=12) | Asacol (N=16)
Nasopharyngitis (Infections and infestations) | 4 | 0 | 1 | 3 | 2 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 3 | 0 | 1 | 3
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 2 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood chloride increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Gamma- glutamyltransferase (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Serum ferritin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.